CLINICAL TRIAL: NCT01830686
Title: Metabolic Effects of Short Term Sugarcane Bagasse Supplementation
Acronym: BROWNIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Daniel Hsia, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: PBRC 13005
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Insulin Resistance
Keywords: Sugarcane bagasse, glucose tolerance, insulin resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sugarcane bagasse (Experimental): 10 subjects will consume food (brownies and cookies) made with 13 g of sugarcane bagasse everyday for 4 weeks
  Interventions: Other: Sugarcane bagasse
- Non-caloric, non-fermentable fiber (Active Comparator): 10 subjects will consume food (brownies and cookies) made with 13 g of non caloric, non-fermentable fiber everyday for 4 weeks
  Interventions: Other: Non-caloric, non-fermentable fiber
- Minimal fiber (Placebo Comparator): 10 subjects will consume food (brownies and cookies) made with 4 g of dietary fiber everyday for 4 weeks
  Interventions: Other: Minimal fiber

INTERVENTIONS:
Other: Sugarcane bagasse — One brownie containing 10 g of sugarcane bagasse and 2 cookies containing 3 g of sugarcane bagasse (total of 13 g of sugarcane bagasse per day)
  Arms: Sugarcane bagasse
Other: Non-caloric, non-fermentable fiber — One brownie containing 10 g of fiber and 2 cookies containing 3 g of fiber (total of 13 g of non-caloric, non-fermentable fiber per day)
  Arms: Non-caloric, non-fermentable fiber
Other: Minimal fiber — One brownie containing 3g of fiber and two cookies containing 1g of fiber (total of 4 g of dietary fiber per day)
  Arms: Minimal fiber

SUMMARY:
The purpose of this study is to help understand the benefits of eating food supplemented with fiber in the form of sugarcane bagasse (the leftover fiber after cane juice is extracted) on glucose metabolism and body weight.

DETAILED DESCRIPTION:
The investigators will employ a double-blind randomized controlled study design with 3 arms such that obese, insulin resistant adults will be randomly selected to receive food made with 1) sugarcane bagasse, 2) non-caloric, non-fermentable fiber, or 3) a similar product with minimal fiber for 4 weeks. The intervention will be in the form of brownies and cookies and will look and taste nearly identical to each other. Caloric value will be constant with all three delivery systems. Subjects will have blood testing and body composition analysis before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18-50 years
* Body Mass Index ≥ 30 kg/m2 (a ratio of weight to height)
* Fasting insulin level >5 µIU/mL, as determined by tests performed during screening

Exclusion Criteria:

* Women who are pregnant
* Past medical history of diabetes
* History of intestinal surgery such as removal of bowel
* History of problems with absorbing food such as celiac disease, inflammatory bowel disease, malabsorption syndrome
* Taking chronic medications for any medical conditions such as diabetes, hypertension, cholesterol, thyroid hormone, etc.
* Any food allergies

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The benefit of sugarcane bagasse on glucose tolerance and insulin resistance in adults with established insulin resistance | 4 weeks
  Participants will be randomly selected to eat food supplemented with either 1) sugarcane bagasse, 2) another type of fiber of equal weight, or 3) minimal fiber. At baseline each eligible subject will have a 3 hour oral glucose tolerance test. Subjects will consume one brownie and two cookies a day for four weeks. At the end of four weeks, the blood tests conducted at baseline will be repeated.

SECONDARY OUTCOMES:
The effect of sugarcane bagasse on body weight/composition | 4 weeks
  At baseline and weekly till the end of the study, weight will be measured. In addition body composition via DXA will be measured at baseline and at the end of the study.

OTHER OUTCOMES:
The effect of sugarcane bagasse on incretin profiles as a mechanism to explain its metabolic effects | 4 Weeks
  At baseline and at the end of the study, glucagon-like peptide-1 and ghrelin levels will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hsia, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No